CLINICAL TRIAL: NCT04111211
Title: Memento-Plus : Long-term Follow-up of Cognitive and Functional Evolutions of Persons With Isolated Cognitive Complaints or Mild Cognitive Deficits
Brief Title: Long-term Follow-up of Cognitive and Functional Evolutions of Persons With Isolated Cognitive Complaints or Mild Cognitive Deficits
Acronym: Memento-Plus
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/16
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; related disorders; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals at high risk of developing Alzheimer's dementia

SUMMARY:
Dementia is a clinical syndrome that is the result of distinct underlying pathologies including Alzheimer's disease (AD). Despite more than two decades of research on prevention and treatment of dementia and aging-related cognitive decline, highly effective preventive and therapeutic strategies remain elusive.

Many features of dementia render it especially challenging. Indeed development of disease occurs insidiously over the course of years or decade. In addition, the causes of dementia and determinants of its severity are likely multi-factorial.

To overcome these challenges and better understand the causes and course of AD and related disorders, long term follow-up studies of persons at high risk of dementia are required including multidimensional and harmonized assessment of risk factors, phenotypes (cognition, neuropsychiatric symptoms, physical health, self rated health) and endophenotypes (blood markers, genetic markers, neuroimaging markers).

This project proposes an extension of the follow-up of Memento participants over 5 to 10 years with of focus on cognitive outcomes and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged over 18 year-old
* Being included in Memento cohort
* Affiliated person or beneficiary of a social security scheme.
* Participants capable of expressing non objection
* Non objection expressed by the tutor for participants under tutorship
* Non objection expressed by the participant assisted by their guardian for participants under guardianship
* Non objection expressed by the trusted person (in accordance with art. L1111-6 of Code de la Santé Publique) for participants without the capacity to express non-objection and who are not under legal protection measure

Exclusion Criteria:

* Expressing opposition to participate in Memento-Plus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from French Research Memory Centers and included in Memento cohort
Sampling Method: Non-Probability Sample
Enrollment: 1028 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Progression to clinical dementia stage according to standardized classifications (DSM-IV for dementia and NINCDS-ADRDA for Alzheimer's disease) | Each 12 months from baseline for 5 years

SECONDARY OUTCOMES:
Mortality | Each 12 months from baseline for 5 years
Loss of autonomy based on functional activity assessment | Each 12 months from baseline for 5 years
Rate of cognitive decline based on change in cognitive performances | Each 12 months from baseline for 5 years
Incidence of neurovascular and cardiovascular events (Stroke and Coronary events) | Each 12 months from baseline for 5 years
Quality of life: EQ-5D (EUROQOL) | Each 12 months from baseline for 5 years
  EQ-5D (EUROQOL) questionnaire Subscales: VAS patient's self-rated health (0=worst, 100=best), mobility, self-care, usual activities, pain/discomfort and anxiety/depression (rated as no problems, slight problems, moderate problems, severe problems and extreme problems)
Incidence of prodromal AD (Pre-symptomatic dementia) | Each 12 months from baseline for 5 years
Incidence of institutionalization | Each 12 months from baseline for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève CHENE, Prof, Principal Investigator — CIC-1401 EC - ISPED - CHU de Bodeaux; Geneviève CHENE, Prof, Study Chair — CIC-1401 EC - ISPED - CHU de Bodeaux; Carole DUFOUIL, Director, Study Director — CIC-1401 EC - ISPED - CHU de Bodeaux
Locations (26):
- France (26):
  - CHU d'Amiens, Amiens
  - AP-HP - CHU Avicenne, Bobigny
  - CHU de Bordeaux - Pellegrin, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHRU de Nice - Institut Claude Pompidou, Nice
  - CHU de Nice - Hôpital de Cimiez, Nice
  - AP-HP - Hôpital BROCA, Paris
  - Ap-Hp La Pitié-Salpêtrière, Paris
  - APHP Groupe Hospitalier Saint Louis Lariboisière Fernand Widal, Paris
  - CHU de Bordeaux, Pessac
  - CHU de Poitiers, Poitiers
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse - Hôpital Purpan, Toulouse
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours
  - Hospice Civil de Lyon, Villeurbanne

IPD SHARING:
Plan to Share IPD: No